CLINICAL TRIAL: NCT02315001
Title: The Physiological Effects of GLP-1 on Haemodynamics During Exercise in Patients With Ischaemic Heart Disease
Brief Title: Liraglutide to Improve corONary Haemodynamics During Exercise streSS
Acronym: LIONESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: RJ112/N131; FS/11/70/28917 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2014-11-10; First posted 2014-12-11 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Ischaemic Heart Disease; Coronary Heart Disease; Chronic Stable Angina
Keywords: Liraglutide; GLP-1; Ischaemic heart disease; Coronary heart disease; Chronic stable angina
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Angina, Stable | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Active Comparator): Week 1 Run-In Phase = 0.6 mg (0.1 ml) Liraglutide once daily via subcutaneous injection
  Week 2 Low-Dose Phase = 1.2 mg (0.2 ml) Liraglutide once daily via subcutaneous injection
  Week 3 High-Dose Phase = 1.8 mg (0.3 ml) Liraglutide once daily via subcutaneous injection
  Interventions: Drug: Liraglutide
- Saline Placebo (Placebo Comparator): Week 1 Run-In Phase = 0.1 ml normal saline once daily via subcutaneous injection
  Week 2 Low-Dose Phase = 0.2 ml normal saline once daily via subcutaneous injection
  Week 3 High-Dose Phase = 0.3 ml normal saline once daily via subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Liraglutide — GLP-1 receptor agonist administered via subcutaneous injection
  Other Names: Victoza
  Arms: Liraglutide
Other: Placebo — Volume-matched normal saline placebo administered via subcutaneous injection
  Arms: Saline Placebo

SUMMARY:
A single-centre double-blind placebo-controlled crossover randomised controlled trial to determine the physiological basis of glucagon-like peptide-1 receptor activation on exercise haemodynamics, as manifest through specific electrophysiological parameters measured by serial exercise stress testing, in those patients with reversible myocardial ischaemia and obstructive coronary artery disease confirmed by a baseline exercise test and coronary angiography respectively.

DETAILED DESCRIPTION:
Glucagon-like peptide-1 (GLP-1), an endogenous incretin hormone, is secreted by the gut in response to enteral nutrition and is responsible primarily for normal glucose homeostasis. There is a defective incretin effect in Type II diabetes mellitus such that meal-stimulated GLP-1 secretion is markedly impaired. However, a continuous infusion of exogenous GLP-1 can result in near normal insulin responses to a glucose load, suggesting preservation of insulinotropic activity. Liraglutide, a synthetic analogue that shares 97% structural homology to native GLP-1, is now a guideline-mandated antidiabetic therapy given as a once-daily subcutaneous injection.

Evidence emerging from animal and latterly human studies suggest GLP-1, independent of its effect on glycemic control and weight loss, may protect the heart from myocardial ischaemia/reperfusion injury and could potentially modulate the metabolic and haemodynamic outcomes of patients with coronary artery disease and left ventricular systolic dysfunction.

The investigators aim to determine whether chronic GLP-1 receptor occupancy has any effect on exercise haemodynamics in patients with known chronic stable angina, evidence of reversible ischaemia on exercise stress testing and angiographic evidence of obstructive coronary artery disease. Each study participant will be randomised to enter either a GLP-1 treatment arm or volume-matched saline placebo arm. Those randomised to GLP-1 will have a week's run-in phase with 0.6 mg Liraglutide followed by a week's course of 1.2 mg Liraglutide. At the end of Week 2, patients in the treatment arm will have their first exercise tolerance test (ETT). They will then be up-titrated to high dose 1.8 mg Liraglutide for another week before performing a Week 3 ETT. Patients in the placebo arm will have matched volume saline injections for the first two weeks before the Week 2 ETT and then another week of saline injections before the Week 3 ETT.

At the end of Week 3 patients will crossover so that those in the GLP-1 treatment arm cross to the placebo arm and vice versa. By incorporating a run-in phase followed by a step-wise increase in Liraglutide therapy over a 3-week period the investigators aim to minimise the occurrence of adverse reactions and also hope to observe a dose-response effect on exercise haemodynamics. The crossover design will allow study participants to effectively act as their own controls.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-80
2. Patients with a recent abnormal exercise tolerance test demonstrating >0.1 mV of planar or down-sloping ST-segment depression.
3. Patients with known coronary artery disease and angiographic evidence of a >70% stenosis in a main epicardial artery, with or without coronary stenoses elsewhere.
4. Patients must be able to walk confidently on a treadmill.
5. Patients must have a normal resting electrocardiogram (ECG) in sinus rhythm without bundle branch aberration or other conduction disturbance.
6. Patients must have normal left ventricular function.

Exclusion Criteria:

1. An abnormal resting ECG including atrial fibrillation, bundle branch aberration or other conduction disturbance.
2. Pre-existing left ventricular systolic dysfunction.
3. Pre-existing ischaemic or non-ischaemic cardiomyopathy.
4. Pre-existing valvular heart disease.
5. Inability to safely negotiate an exercise treadmill.
6. Type I diabetes mellitus.
7. Type II diabetes mellitus taking oral or subcutaneous anti diabetic therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in rate pressure product at 0.1 mV ST-segment depression | Following consecutive exercise treadmill tests performed at Week 2, Week3, Week 5 and Week 6 of a 6-week study protocol
Change in degree of ST-segment depression at peak exercise | Following consecutive exercise treadmill tests performed at Week 2, Week3, Week 5 and Week 6 of a 6-week study protocol

SECONDARY OUTCOMES:
Change in total exercise duration | Following consecutive exercise treadmill tests performed at Week 2, Week3, Week 5 and Week 6 of a 6-week study protocol
Change in time to 0.1 mV ST-segment depression | Following consecutive exercise treadmill tests performed at Week 2, Week3, Week 5 and Week 6 of a 6-week study protocol
Change in recovery time to 0.05 mV ST-segment depression | Following consecutive exercise treadmill tests performed at Week 2, Week3, Week 5 and Week 6 of a 6-week study protocol
Evidence of hypoglycaemia | During 6-week study protocol
  Monitored via twice daily home glucose monitoring and once weekly random serum glucose measurements
Evidence of renal dysfunction | During 6-week study protocol
  Monitored via once weekly measurement of serum creatinine, electrolytes and estimated glomerular filtration rate
Evidence of acute pancreatitis | During 6-week study protocol
  Monitored via once weekly measurement of serum amylase along with telephone and once weekly face-to-face interviews
Change in time to maximum ST-segment depression | Following consecutive exercise treadmill tests performed at Week 2, Week3, Week 5 and Week 6 of a 6-week study protocol

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marber, PhD FRCP, Principal Investigator — King's College London; Simon Redwood, MD FRCP, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, Greater London, United Kingdom

REFERENCES:
- [Background] Myat A, Arri S, Bhatt DL, Gersh BJ, Redwood SR, Marber MS. Design and rationale for the randomised, double-blinded, placebo-controlled Liraglutide to Improve corONary haemodynamics during Exercise streSS (LIONESS) crossover study. Cardiovasc Diabetol. 2015 Feb 19;14:27. doi: 10.1186/s12933-015-0193-4. PMID 25848859
- [Derived] Myat A, Redwood SR, Arri S, Gersh BJ, Bhatt DL, Marber MS. Liraglutide to Improve corONary haemodynamics during Exercise streSS (LIONESS): a double-blind randomised placebo-controlled crossover trial. Diabetol Metab Syndr. 2021 Feb 12;13(1):17. doi: 10.1186/s13098-021-00635-6. PMID 33579317
- See also: Trial rationale and protocol — http://www.cardiab.com/content/14/1/27